CLINICAL TRIAL: NCT03029143
Title: A Phase 4 Open-Label Study to Evaluate Vedolizumab IV Dose Optimization on Treatment Outcomes In Nonresponders With Moderately to Severely Active Ulcerative Colitis (ENTERPRET)
Brief Title: Vedolizumab Intravenous (IV) Dose Optimization in Ulcerative Colitis
Acronym: ENTERPRET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4014; U1111-1183-0451 (Other: WHO)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Colitis, Ulcerative
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lead-in Period: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg intravenous (IV) infusion once at Day 1 and at Week 2. Participants who were non-responders based on partial Mayo score at Week 6 and who had high vedolizumab clearance (>0.14 L/day) at Week 5 were eligible for Randomized Treatment Period (RTP). Participants who were responders (Lead-In Failures) entered the 18-week follow-up period and discontinued the study.
  Interventions: Drug: Vedolizumab IV
- Randomized Treatment Period (RTP): Standard Treatment Arm (Experimental): Following Lead-in Period, participants received vedolizumab 300 mg, IV infusion, once every 8 weeks (Q8W) at Weeks 6, 14 and 22 as standard treatment plus 18 weeks follow-up.
  Interventions: Drug: Vedolizumab IV
- RTP: Dose Optimized Arm (Experimental): Following Lead-in Period, participants received vedolizumab 600 mg, IV infusion at Week 6, followed by Regimen A: vedolizumab 300 mg once in every 4 weeks (Q4W) thereafter (Weeks 10, 14, 18, 22 and 26) plus 18 weeks follow-up, or Regimen B: vedolizumab 600 mg, IV infusion Q4W (Weeks 10, 14, 18, 22 and 26) plus 18 weeks follow-up based on drug clearance.
  Interventions: Drug: Vedolizumab IV

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab intravenous infusion.
  Other Names: Entyvio; MLN0002

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of vedolizumab intravenous (IV) dose optimization on mucosal healing compared with the standard vedolizumab IV dosing regimen over a 30 week treatment period in participants with moderately to severely active ulcerative colitis (UC) and high vedolizumab clearance, based on a Week 5 predefined serum vedolizumab concentration threshold less than (<) 50 microgram per milliliter (microg/mL) and who are Week 6 non-responders based on partial Mayo score.

DETAILED DESCRIPTION:
The drug being tested in this study is called Vedolizumab. Vedolizumab will be administered as an IV infusion. It is being tested in this study with new doses. This study will investigate the efficacy and safety of dose optimization of vedolizumab IV, compared with standard dosing of vedolizumab IV, over a 30-week treatment period.

The study will enroll approximately 250 moderately to severely active subjects with UC in order to randomize approximately 100 non-responder subjects with high vedolizumab drug clearance. Subjects will receive induction therapy of vedolizumab IV 300 mg on Day 1 and Week 2 (Lead-in Period). At Week 5, serum vedolizumab concentration will be measured. At Week 6, subjects will be assessed for clinical response based on partial Mayo score.

Results of both Week 5 vedolizumab concentration and Week 6 clinical response will determine the treatment pathway. Those who are non-responders based on partial Mayo score at Week 6 and who are assessed as having high vedolizumab clearance, based on a predefined Week 5 serum vedolizumab concentration threshold (<50 microg/mL) will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Vedolizumab IV Standard Treatment
* Vedolizumab IV Dose Optimized

All randomized subjects will receive vedolizumab IV either 300 mg or 600 mg every 4 or 8 weeks.

This multi-center trial will be conducted in United States of America and Canada. The overall time to participate in this study is 56 weeks. Subjects will make multiple visits to the clinic, and will be contacted by telephone, 6 months after last dose of study drug for a long term follow-up safety survey.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of UC established at least 1 month prior to Screening by clinical and endoscopic evidence and corroborated by a histopathology report.
2. Has moderately to severely active UC as determined by a complete Mayo score of 6 to 12 with an endoscopic subscore ≥2 within 28 days prior to enrollment.
3. Has evidence of UC proximal to the rectum (≥15 cm of involved colon) prior to start of vedolizumab IV dosing.
4. Has been determined to be suitable for vedolizumab IV for routine management of UC by their physician.
5. Has a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factor must be up-to-date on colorectal cancer surveillance (may be performed during screening).
6. Has demonstrated an inadequate response with, lost response to, or intolerance of at least 1 of the following agents: immunomodulators, corticosteroids, or tumor necrosis factor-alpha (TNF-α) antagonists. Subject who are naive to TNF-α antagonist therapy or who have previously failed TNF-α antagonist therapy (including primary and secondary non-responders or intolerant) may be included.

   Week 6 Randomized Treatment Period Inclusion Criteria
7. Following Lead-in Period, the subject is assessed as having high vedolizumab drug clearance based on a predefined Week 5 serum vedolizumab concentration threshold (<50 microg/mL).
8. Following Lead-in Period, the subject is a non-responder based on partial Mayo score at Week 6.

Exclusion Criteria:

1. Has clinical evidence of abdominal abscess or toxic megacolon at the Screening Visit.
2. Has had an extensive colonic resection, subtotal or total colectomy.
3. Has had ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
4. Has a diagnosis of Crohn's colitis or indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
5. Has received any of the following for the treatment of underlying disease within 30 days of screening:

   1. Non-biologic therapies (eg. cyclosporine, tacrolimus, thalidomide)
   2. An approved non-biologic therapy in an investigational protocol.
6. Has received any investigational or approved biologic or biosimilar agent within 60 days or 5 half-lives prior to screening (whichever is longer).
7. Has previously had prior exposure to approved or investigational anti-integrin antibodies (e.g. natalizumab, efalizumab, etrolizumab, AMG-181, anti-MAdCAM-1 antibodies or rituximab).
8. Has previously received approved or investigational vedolizumab.
9. The subject currently requires or is anticipated to require surgical intervention for UC during the study.
10. Has history or evidence of adenomatous colonic polyps that have not been removed, or colonic mucosal dysplasia.
11. Has any evidence of an active infection during Screening (eg, sepsis, cytomegalovirus, or listeriosis).
12. Has a clinically significant infection (eg, pneumonia, pyelonephritis) within 30 days prior to screening, or ongoing chronic infection.
13. Has evidence of active C. difficile as evidenced by positive C. difficile toxin or is having treatment for C. difficile infection or other intestinal pathogens during Screening.
14. Has a known history of infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or chronic HBV (HBV immune subjects (ie, being hepatitis B surface antigen [HBsAg] negative and hepatitis B antibody positive) may, however, be included), or hepatitis C virus (HCV) infection. Subjects with documented successful treatment of HCV with sustained virological response (SVR) at 26 weeks can be enrolled.
15. Has active or latent tuberculosis (TB), as evidenced by the following:

    a. A diagnostic TB test performed within 30 days of screening or during the Screening Period that is positive, defined as: i. Positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, OR ii. A TB skin test reaction ≥ 5 mm OR, b. Chest X-ray within 3 months of screening that is suspicious for pulmonary TB, and a positive or 2 successive indeterminate QuantiFERON tests within 30 days prior to Screening or during the Screening Period.
16. Has any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency, HIV infection, organ transplantation).
17. Has any live vaccination within 30 days prior to Screening or is planning to receive any live vaccination during participation in the study.
18. Has used a topical (rectal) treatment with (5-ASA) or corticosteroid enemas/suppositories within 2 weeks prior to Screening.
19. Has a history of hypersensitivity or allergies to vedolizumab IV or its components.
20. Has received total parenteral nutrition (TPN) or albumin in the last 30 days prior to screening.
21. Has any unstable or uncontrolled cardiovascular disorder, heart failure moderate to severe (New York Class Association III or IV), any pulmonary, hepatic, renal, GI, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise subject safety.
22. Has had a surgical procedure requiring general anesthesia within 30 days prior to screening or is planning to undergo major surgery during the study period.
23. Has a history of malignancy, except for the following: adequately-treated non-metastatic basal cell skin cancer; squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to Screening; and history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to screening. Subjects with remote history of malignancy (eg, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case by-case basis prior to Screening.
24. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, demyelinating, or neurodegenerative disease.
25. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist during Screening or prior to the administration of the first dose of study drug on Day 1.
26. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (49):
- United States (44):
  - Advanced Clinical Therapeutics, LLC, Tucson, Arizona
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Care Access Research LLC, San Pablo, California
  - Care Access Research, San Pablo, San Pablo, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Gastro Florida, Clearwater, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Wellness Clinical Research, LLC, Hialeah, Florida
  - Center for Advanced Gastro, Maitland, Florida
  - Center for Interventional Endo, Orlando, Florida
  - BRCR Medical Center, Inc., Pembroke Pines, Florida
  - Gastro Florida, Tampa, Florida
  - Atlanta Gastroenterology Specialists, PC, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, Decatur, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - NorthShore University HealthSystem, Evanston, Illinois
  - Aquiant Research, New Albany, Indiana
  - Iowa Digestive disease center, Clive, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - 4940 Eastern Ave A building, Baltimore, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Weill Cornell Medical College, New York, New York
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Gastroenterology Associates PA, Greenville, South Carolina
  - Midwest Medical Care, Sioux Falls, South Dakota
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Ygenics, Decatur, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Digestive Disease Consultants, Keller, Texas
  - DHAT Research Institute, Richardson, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - BaylorScott&White Research Institute, Temple, Texas
  - GI Liver Research LLC, Webster, Texas
  - Gastroenterology Associates of Northern Virginia, Ltd., Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Canada (5):
  - PerCuro Clinical Research Ltd., Victoria, British Colombia
  - LHSC - University Hospital, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Taunton Surgical Centre, Oshawa, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Jairath V, Yarur A, Osterman MT, James A, Balma D, Mehrotra S, Yang L, Yajnik V, Qasim Khan RM. ENTERPRET: A Randomized Controlled Trial of Vedolizumab Dose Optimization in Patients With Ulcerative Colitis Who Have Early Nonresponse. Clin Gastroenterol Hepatol. 2024 May;22(5):1077-1086.e13. doi: 10.1016/j.cgh.2023.10.029. Epub 2023 Nov 10. PMID 37951560
- See also: To obtain more information on the study, click on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60394db2bf003ab4a241?idFilter=%5B%22Vedolizumab-4014%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with ulcerative colitis (UC) took part in the study at 90 investigative sites in the United States and Canada from 29 March 2017 to 16 October 2020.
Pre-assignment Details: Participants with UC enrolled in Lead-in Period received vedolizumab 300 mg at Day 1 and Week 2. At Week 5, participants were assessed for clearance and at Week 6 for clinical response per partial Mayo Score. The non-responders were randomized to receive optimized treatment (Regimen A or B, dose decided by vedolizumab clearance) or standard vedolizumab treatment. The responders or participants with low vedolizumab clearance received vedolizumab 300 mg at Week 6 plus 18-week follow-up.
Groups:
- Lead-in Period: Vedolizumab 300 mg: Vedolizumab 300 mg intravenous (IV) infusion once at Day 1 and at Week 2. Participants were then assessed to estimate the vedolizumab clearance at Week 5 and response at Week 6.
- RTP: Dose Optimized Arm: Following Lead-in Period participants received vedolizumab 600 mg, IV infusion at Week 6, followed by Regimen A: vedolizumab 300 mg once in every 4 weeks (Q4W) thereafter (Weeks 10, 14, 18, 22 and 26) plus 18 weeks follow-up, or Regimen B: vedolizumab 600 mg, IV infusion Q4W (Weeks 6, 10, 14, 18, 22 and 26) plus 18 weeks follow-up based on drug clearance.
Period: Lead-in Period (6 Weeks)
Arm/Group | Lead-in Period: Vedolizumab 300 mg | Randomized Treatment Period (RTP): Standard Treatment Arm | RTP: Dose Optimized Arm
Started | 278 | 0 | 0
Completed (Completed = Participants who were eligible for randomization or randomized in error; Not completed = Participants who were Lead-In Failure. One participant was randomized to Randomized Treatment Period: Standard Treatment Arm, but was not treated and was thus presented in the Lead-in failure vedolizumab arm for the Safety Analysis Set (N=170).) | 109 | 0 | 0
Not Completed | 169 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 8 | 0 | 0
Not completed — Significant Protocol Deviation | 12 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 6 | 0 | 0
Not completed — Randomized but not Treated | 142 | 0 | 0
Period: Randomized Treatment Period (24 Weeks)
Arm/Group | Lead-in Period: Vedolizumab 300 mg | Randomized Treatment Period (RTP): Standard Treatment Arm | RTP: Dose Optimized Arm
Started | 0 | 54 | 55
Not Treated Post Randomization | 0 | 1 (One participant was randomized to Randomized Treatment Period: Standard Treatment Arm, but was not treated and was thus included in the Lead-in failure vedolizumab arm for the Safety Analysis Set (N=170).) | 0
Safety Population (Safety Analysis Set included all participants who were enrolled and received at least one dose of study medication.) | 0 | 53 | 55 (Regimen A = 28 Regimen B = 27)
Completed | 0 | 31 | 31
Not Completed | 0 | 23 | 24
Not completed — Pretreatment Event/Adverse Event | 0 | 3 | 9
Not completed — Significant Protocol Deviation | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Voluntary Withdrawal | 0 | 10 | 1
Not completed — Lack of Efficacy | 0 | 6 | 7
Not completed — Reason not Specified | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set Included all participants who were enrolled and received at least one dose of study medication.
Groups:
- Lead-in Period: Vedolizumab 300 mg: Vedolizumab 300 mg intravenous (IV) infusion once at Day 1 and at Week 2 . Participants were then assessed to estimate the vedolizumab clearance at Week 5 and response at Week 6.
Arm/Group | Lead-in Period: Vedolizumab 300 mg
Number analyzed (Participants) | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34
  Not Hispanic or Latino | 244
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 28
  White | 228
  More than one race | 2
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 171.5 (9.39)
Weight [Mean (Standard Deviation); unit: kg] | 80.41 (20.112)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight (kg)/[height (m)^2].
  kg/m^2 | 27.24 (5.942)
Smoking Classification [Count of Participants; unit: Participants]
  Participant has never smoked | 179
  Participant is a current smoker | 12
  Participant is an ex-smoker | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Mucosal Healing at Week 30
Description: Mucosal healing is defined as Mayo endoscopic subscore <=1 point. Mayo score was used in clinical trials to assess UC disease activity. It consisted of 4 disease activity variables (stool frequency, rectal bleeding, findings on sigmoidoscopy and physician's global assessment), each scored on a scale of 0 to 3, where 0 normal condition and 3 = severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.
Time Frame: Week 30
Population: Full Analysis Set included all participants who were randomized and received at least one dose of study medication post-randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RTP: Standard Treatment Arm: Following Lead-in Period participants received vedolizumab 300 mg, IV infusion, once at Weeks 6, 14 and 22 [every 8 weeks (Q8W)] as standard treatment plus 18 weeks follow-up.
Arm/Group | RTP: Standard Treatment Arm | RTP: Dose Optimized Arm
Number analyzed (Participants) | 53 | 55
percentage of participants | 18.9 [9.4 to 32.0] | 14.5 [6.5 to 26.7]
Statistical Analysis 1: Comparison: RTP: Standard Treatment Arm vs RTP: Dose Optimized Arm; Test type: Other; p = 0.401, Chi-squared; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.2 to 1.8]; Chi-squared test was used to estimate P-value from the logistic regression model where Endoscopic Mucosal Healing was the response variable and Treatment and TNF stratification were factors. Baseline complete Mayo Score and natural logarithm of trough concentration at week 6 were covariates

2. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 30
Description: Clinical remission is defined as a complete Mayo score of ≤2 points and no individual subscore >1 point at Week 30. Mayo score was used in clinical trials to assess UC disease activity. It consisted of 4 disease activity variables (stool frequency, rectal bleeding, findings on sigmoidoscopy and physician's global assessment), each scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.
Time Frame: Week 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTP: Standard Treatment Arm | RTP: Dose Optimized Arm
Number analyzed (Participants) | 53 | 55
percentage of participants | 9.4 [3.1 to 20.7] | 9.1 [3.0 to 20.0]
Statistical Analysis 1: Comparison: RTP: Standard Treatment Arm vs RTP: Dose Optimized Arm; Test type: Other; p = 0.943, CMH Chi-square test; Adjusted risk difference = -0.4, 95% CI 2-sided [-11.4 to 10.6]; Cochran-Mantel-Haenszel (CMH) chi-square test was stratified by TNF antagonist status

3. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 30
Description: Clinical response is defined as a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline (Day 1) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point, at Week 30. Mayo score was used in clinical trials to assess UC disease activity. It consisted of 4 disease activity variables (stool frequency, rectal bleeding, findings on sigmoidoscopy and physician's global assessment), each scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.
Time Frame: Week 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | RTP: Standard Treatment Arm | RTP: Dose Optimized Arm
Number analyzed (Participants) | 53 | 55
percentage of particpants | 32.1 [19.9 to 46.3] | 30.9 [19.1 to 44.8]
Statistical Analysis 1: Comparison: RTP: Standard Treatment Arm vs RTP: Dose Optimized Arm; Test type: Other; p = 0.893, CMH Chi-square test; Adjusted risk difference = -1.2, 95% CI 2-sided [-18.7 to 16.3]; Cochran-Mantel-Haenszel (CMH) chi-square test was stratified by TNF antagonist status

4. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 14
Description: Clinical response is defined as A reduction in partial Mayo score of ≥2 points and ≥25% from Baseline (Day 1) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. Mayo score was used in clinical trials to assess UC disease activity. A composite index of 3 disease activity variables (stool frequency, rectal bleeding, and physician's global assessment), each scored on a scale from 0 to 3 with total partial Mayo score ranging from 0 to 9 (higher scores indicate greater disease activity). Partial Mayo score is calculated analogously to the complete Mayo score but excludes the sigmoidoscopy subscore.
Time Frame: Week 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTP: Standard Treatment Arm | RTP: Dose Optimized Arm
Number analyzed (Participants) | 53 | 55
percentage of participants | 34.0 [21.5 to 48.3] | 40.0 [27.0 to 54.1]
Statistical Analysis 1: Comparison: RTP: Standard Treatment Arm vs RTP: Dose Optimized Arm; Test type: Other; p = 0.525, CMH Chi-square test; Adjusted risk difference = 6.0, 95% CI 2-sided [-12.4 to 24.3]; Cochran-Mantel-Haenszel (CMH) chi-square test was stratified by TNF antagonist status

5. Secondary Outcome: Percentage of Participants Achieving Corticosteroid-Free Remission
Description: Participants using oral corticosteroids at Baseline who have discontinued corticosteroids and are in clinical remission. Mayo score was used in clinical trials to assess UC disease activity. Clinical Remission is defined as a complete Mayo score of <=2 points and no individual subscore >1 point at Week 30. It consisted of 4 disease activity variables (stool frequency, rectal bleeding, findings on sigmoidoscopy and physician's global assessment), each scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.
Time Frame: Week 30
Population: Full Analysis Set included all participants who were randomized and received at least one dose of study medication post-randomization. Overall number analyzed are the participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTP: Standard Treatment Arm | RTP: Dose Optimized Arm
Number analyzed (Participants) | 14 | 21
percentage of participants | 21.4 [4.7 to 50.8] | 14.3 [3.0 to 36.3]
Statistical Analysis 1: Comparison: RTP: Standard Treatment Arm vs RTP: Dose Optimized Arm; Test type: Other; p = 0.623, CMH Chi-square test; Adjusted risk difference = -6.6, 95% CI 2-sided [-34.0 to 20.8]; Cochran-Mantel-Haenszel (CMH) chi-square test was stratified by TNF antagonist status

6. Secondary Outcome: Percentage of Participants Achieving Durable Clinical Response
Description: A clinical response (based on partial Mayo score), which is defined as a reduction in partial Mayo score of ≥2 points and ≥25% from Baseline with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at Weeks 14 and 30. Mayo score was used in clinical trials to assess UC disease activity. A composite index of 3 disease activity variables (stool frequency, rectal bleeding, and physician's global assessment), each scored on a scale from 0 to 3 with total partial Mayo score ranging from 0 to 9 (higher scores indicate greater disease activity). Partial Mayo score is calculated analogously to the complete Mayo score but excludes the sigmoidoscopy subscore. Percentage of participants with durable clinical response, clinical response achieved at both Weeks 14 and 30 are reported.
Time Frame: Weeks 14 and 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTP: Standard Treatment Arm | RTP: Dose Optimized Arm
Number analyzed (Participants) | 53 | 55
percentage of participants | 22.6 [12.3 to 36.2] | 30.9 [19.1 to 44.8]
Statistical Analysis 1: Comparison: RTP: Standard Treatment Arm vs RTP: Dose Optimized Arm; Test type: Superiority; p = 0.344, CMH Chi-square test; Adjusted risk difference = 8.1, 95% CI 2-sided [-8.5 to 24.7]; Cochran-Mantel-Haenszel (CMH) chi-square test was stratified by TNF antagonist status

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 18 weeks after the last dose (approximately 44 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Data is reported for Safety Analysis Set, as per the treatment received throughout the study. Data for adverse events for Regimen A and B are reported per dose.
Groups:
- Lead-in Period: Vedolizumab 300 mg intravenous (IV) infusion once at Day 1 and at Week 2.
- Lead-in Failure Follow-up Period: Following Lead in Period, participants who were responders at Week 6 or had normal-to-low vedolizumab clearance at Week 5 were not eligible for randomization and received vedolizumab 300 mg IV infusion at Week 6 plus 18 weeks follow-up.
- RTP: Standard Treatment Arm: Following Lead-in Period, participants received vedolizumab 300 mg, IV infusion, once at Weeks 6, 14 and 22 [every 8 weeks (Q8W)] as standard treatment plus 18 weeks follow-up.
- RTP: VDZ Dose Optimization: Regimen A: Following Lead-in Period, participants received vedolizumab 600 mg at Week 6 and 300 mg IV infusion once every 4 weeks up to Week 26 in regimen A plus 18 weeks follow-up.
- RTP: VDZ Dose Optimization: Regimen B: Following Lead-in Period, participants received vedolizumab 600 mg at Week 6 followed by vedolizumab 600 mg once every 4 weeks up to Week 26 in regimen B plus 18 weeks follow-up.
Arm/Group | Lead-in Period | Lead-in Failure Follow-up Period | RTP: Standard Treatment Arm | RTP: VDZ Dose Optimization: Regimen A | RTP: VDZ Dose Optimization: Regimen B
All-Cause Mortality (participants affected / at risk) | 1/278 | 0/170 | 0/53 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 12/278 | 1/170 | 4/53 | 4/28 | 1/27
Other Adverse Events (participants affected / at risk) | 10/278 | 4/170 | 9/53 | 12/28 | 9/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Period (N=278) | Lead-in Failure Follow-up Period (N=170) | RTP: Standard Treatment Arm (N=53) | RTP: VDZ Dose Optimization: Regimen A (N=28) | RTP: VDZ Dose Optimization: Regimen B (N=27)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Benign familial haematuria (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 7 | 1 | 2 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Period (N=278) | Lead-in Failure Follow-up Period (N=170) | RTP: Standard Treatment Arm (N=53) | RTP: VDZ Dose Optimization: Regimen A (N=28) | RTP: VDZ Dose Optimization: Regimen B (N=27)
Headache (Nervous system disorders) | 8 | 1 | 1 | 3 | 2
Colitis ulcerative (Gastrointestinal disorders) | 2 | 2 | 4 | 0 | 3
C-reactive protein increased (Investigations) | 1 | 1 | 3 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03029143/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03029143/SAP_001.pdf